CLINICAL TRIAL: NCT03449771
Title: Screening of Psychoactive Substances Use and Anxio-depressive Disorders in Consultation for HIV Pre-exposure Prophylaxis
Brief Title: PrEP and Consumptions
Acronym: PrEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion of the last patient
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9878
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Psychoactive Substance Use; Mood Disorders
Keywords: HIV; Pre-exposure prophylaxis; Recreational drugs; Chemsex; Mental disorders
MeSH Terms: conditions — Mood Disorders; Chemsex; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): To estimate the acceptability and the impact on the management of a systematic identification of the use of psychoactive substances and / or anxio-depressive disorders by self-questionnaire.
  Interventions: Other: self-administered questionnaire

INTERVENTIONS:
Other: self-administered questionnaire — The newsletter and a self-questionnaire will be systematically given in the waiting room to any PrEP consultant to evaluate the consumption of psychoactive substances (ASSIST questionnaire) and to identify anxio-depressive disorders (HAD questionnaire - Hospital Anxiety and Depression). scale).

SUMMARY:
HIV pre-exposure prophylaxis (PrEP) with Truvada®, a combination of two antiretrovirals (tenofovir & emtricitabine) is a prevention strategy for HIV-negative people at high risk of acquiring HIV. PrEP has thus been integrated as a new tool to significantly reduce the risk of HIV infection, especially among men who have sex with men (MSM). Since its introduction, an increase in sexually transmitted infections (STIs) has been observed, particularly in relation to the use of psychoactive substances in a sexual context (Chemsex).

In this context, the description and evaluation of these practices seem necessary, as well as the impact on the risk of addiction and mental health.

DETAILED DESCRIPTION:
Interventional, multi-center pilot study, including all subjects aged 18 years or older presenting in consultation for a PrEP renewal.

The newsletter and a self-questionnaire will be systematically given in the waiting room to any PrEP consultant to evaluate the consumption of psychoactive substances (ASSIST questionnaire) and to identify anxio-depressive disorders (HAD questionnaire - Hospital Anxiety and Depression). scale). After consent, the answers will be discussed with the doctor during the consultation for appropriate care, including a referral to a psychiatrist and / or addictologist if necessary.

The duration of the inclusions will be 6 months and the number of patients to include is 250.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged over 18,
* Subject seen in consultation in one of the centers of the study for a renewal of the Prep
* Subject having agreed to participate in the study

Exclusion Criteria:

* Subject not speaking French / illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-11-03 (Actual)

PRIMARY OUTCOMES:
Estimate the acceptability and the impact on the management of a systematic identification of the use of psychoactive substances and / or anxio-depressive disorders by self-questionnaire in PrEP consultants | 1 year after the study start date

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Hospital of Alès, Alès
  - Uh Montpellier, Montpellier
  - CEGIDD, Nîmes
  - UH NIMES, Nîmes
  - Hospital of Perpignan, Perpignan

IPD SHARING:
Plan to Share IPD: No